CLINICAL TRIAL: NCT00623207
Title: Safety and Feasibility of Atropine Added During Treadmill Stress Testing in Patients With Chronotropic Incompetence or Poor Exercise Capacity.
Brief Title: Use of Atropine in Tredmill Stress Testing
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Mohamed Jabaren, MD, HaEmek Medical Center, Israel
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 07-0139 EMC
Record Dates: First submitted 2008-02-14; First posted 2008-02-25 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2015-07

CONDITIONS: Chest Pain
Keywords: Chest Pain Low work Capacity Rate Incompetence
MeSH Terms: conditions — Chest Pain | interventions — Atropine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): Pateints who achieve target haert rate or conclusive test will not be given Atropine
  Interventions: Drug: Atropine
- 2 (Active Comparator): Patients who won't achieve tarhet heart rate or conclusive results will be given Atropine
  Interventions: Drug: Atropine

INTERVENTIONS:
Drug: Atropine — I.V Atropine 0.5mg up to 2 mg

SUMMARY:
The aim of this study is to evaluate the Safety and feasibility of atropine added during treadmill stress testing in patients with chronotropic incompetence or poor exercise capacity.

Our hypothesis is that we can increase heart rate by using atropin in these patients, so we will achieve more conclusive results.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chest pain without evidence of ischemia eligible for exercise test.
* Age> 18 years old

Exclusion Criteria:

Absolute:

* Patients with LBBB
* Unstable Angina
* Recent Myocardial Infarction
* Un controlled Arrythmia
* Congestive heart faliure
* Severe symptomatic valvular heart disease
* Acute Pulmonary Embolism
* Acute perimyocarditis
* Acute aortic dissection

Relative:

* Lt main stenosis
* Severe hypertention (Systolic> 200 mmHg; Diastolic > 100 mmHg)
* Cardiomyopathy
* Obstructiove abnormalities
* Psychiatric disorders
* High degree AV Block

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2007-12; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
1- To characterize patients who can't achieve target heart rate at treadmill exercise test.2- To evaluate atropine added during treadmill stress testing in order to increase heart rate and achieave conclusive test. | 1 yaer

CONTACTS AND LOCATIONS:
Locations (1):
- Heart Institute, Ha'Emek Medical Center, Afula, Afula, Israel